CLINICAL TRIAL: NCT02678858
Title: Efficacy of "Integrated Social Cognitive and Behavioral Skills Therapy" (ISST) in Improving Functional Outcome in Schizophrenia
Brief Title: Efficacy of ISST in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: University Hospital, Bonn (Other); University Hospital of Cologne (Other); University Hospital Tuebingen (Other); Zentralinstitut für Seelische Gesundheit Mannheim (Other); University of Cologne (Other); Rheinhessen-Fachklinik Alzey (Other); Vivantes Klinikum am Urban (Unknown)
Responsible Party: Principal Investigator, Wolfgang Wölwer, Prof. Dr. phil., Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISST2015
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia
Keywords: social cognition; social skills; cognitive remediation; functional outcome; treatment adherence
MeSH Terms: conditions — Schizophrenia; Social Skills; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated Social Cognitive and Behavioral Skills Therapy (Experimental): The Integrated Social Cognitive and Behavioral Skills Therapy (ISST) shall target expressive and interactional behavior skills together with those social cognitive domains (facial and prosodic affect recognition, social perception, theory-of-mind) known to be most impaired (Savla, 2012) and most closely associated with functional outcome (Fett, 2012) in schizophrenia.
  Interventions: Behavioral: Integrated Social Cognitive and Behavioral Skills Therapy
- Neurocognitive Remediation Therapy (Active Comparator): The Neurocognitive Remediation Therapy (NCRT) shall target impairments in attention, memory, and executive functions as an active comparator to the ISST.
  Interventions: Behavioral: Neurocognitive Remediation Therapy

INTERVENTIONS:
Behavioral: Integrated Social Cognitive and Behavioral Skills Therapy — The Integrated Social Cognitive and Behavioral Skills Therapy (ISST) is a newly developed treatment program. It is based on the Training of Affect Recognition (Wölwer et al. 2005) and common social skills trainings, which are combined in an integrated rather than a sequenced manner. ISST uses both repeated practice and strategy-based training, and consists of 12 individual sessions, 5 group sessions and 1 individual final session over a period of 6 months.
  Other Names: ISST
  Arms: Integrated Social Cognitive and Behavioral Skills Therapy
Behavioral: Neurocognitive Remediation Therapy — The Neurocognitive Remediation Program (NCRT) is based on a neurocognitive training already used as active control condition in our earlier studies (Wölwer et al. 2005, Klingberg et al. 2011). The present version of NCRT is matched in dose, mode and scheme of application to the ISST, but differs from the ISST regarding targeted cognitive domains and preferred training strategy (predominantly drill and practice based). The NCRT provides the same amount of group interaction and companionship as well as the same amount of guided community activity as in the ISST, but is structured in such a way that interactional behavior is secondary (e.g. by competition-like tasks rather than cooperative tasks). Thus therapeutic attention and commitment are held constant across study conditions.
  Other Names: NCRT
  Arms: Neurocognitive Remediation Therapy

SUMMARY:
The ISST study investigates whether integrated social cognitive remediation and social behavioral skills therapy is more efficacious in improving functional outcome and treatment adherence than an active control treatment comprising drill-and-practice oriented neurocognitive remediation.

DETAILED DESCRIPTION:
Deficits in social functioning are a defining, very burdening feature of schizophrenia precluding patients from participating in a satisfying life. Traditional drug and psychosocial therapy and available specific treatment strategies that directly target single key determinants of functional outcome like neurocognition, social cognition, and social behavioral skills have produced only moderate effects leaving an urgent need for further optimization. The present trial aims to more efficaciously improve functional outcome by integrating social behavioral and social cognitive treatment strategies. Six months of "Integrated Social Cognitive and Behavioral Skills Therapy (ISST)" will be compared with "Neurocognitive Remediation Therapy (NCRT)" as active control condition in a randomized multicenter clinical trial using a two group pre-post design with 2x90 patients in the remitted early phase of schizophrenia. Beyond "all-cause-discontinuation" as common primary outcome of all clinical trials of the ESPRIT-consortium, measures of functional outcome and subjective quality of life, patient experience as well as neurocognitive, social-cognitive and social behavioral measures will be assessed at baseline (V0), after completion of treatment (V6), and after 6 months follow-up (V12). ISST is expected to reduce the one-year discontinuation rate by 20% compared with NCRT, and to be superior in functional outcome measures by an effect size of at least d=0.42.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* DSM-IV-TR diagnosis of schizophrenia (295.10-30, 295.90)
* PANSS at baseline: total score ≤ 75
* Proficiency in German language.

Exclusion Criteria:

* Lack of accountability
* Positive urine drug-screening for illicit drugs at screening (except cannabinoids and benzodiazepines)
* Serious suicidal risk at screening visit
* Other relevant axis 1-diagnoses according to diagnostic interview (MINI);
* Other relevant neurological or somatic disorders
* Verbal IQ<80 (MWT-B)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2016-03; Primary Completion 2021-02 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
All Cause Discontinuation | 6 months, 12 months
  All Cause Discontinuation is defined as 1) not keeping appointments to treatment or diagnostic sessions as scheduled for more than 6 weeks and/or (2) not being traceable despite extensive efforts by the intervention team to reengage the patient throughout the entire intended treatment period and/or (3) withdrawal of consent by the patient (4) rater induced discontinuation of the study treatment (eg. for safety criteria) (5) not taking psychotropic drugs as prescribed for more than 14 consecutive days and/or (6) relevant worsening of symptoms.

SECONDARY OUTCOMES:
Treatment Adherence 1 | 6 months, 12 months
  SES (Service Engagement Scale, Tait, Birchwood & Trower 2002)
Treatment Adherence 2 | 6 months, 12 months
  DAI-10 (Drug Attitude Scale, Goodstadt et al. 1978)
Treatment Adherence 3 | 6 months, 12 months
  PATHEV (Psychotherapy Attitude Scale, Schulte 2005)
Psychosocial Functioning 1 | 6 months, 12 months
  FROGS (Functional Remission of General Schizophrenia, Lorca et al. 2009)
Psychosocial Functioning 2 | 6 months, 12 months
  UPSA-Brief (University of California Performance Based Skills Assessment, Mausbach et al. 2007)
WHOQUOL-Bref (Quality of Life) | 6 months, 12 months
  WHOQUOL-BREF (World Health Organization Quality of Life, WHO 1996)
Neurocognitive Performance (verbal memory) | 6 months, 12 months
  VLMT (verbal learning and memory test, Helmstaedter, Lendt & Lux 2001
Neurocognitive Performance (working memory) | 6 months, 12 months
  DSF, DSB (digit sequencing forward/backward, Wechsler 1981)
Neurocognitive Performance (processing speed 1) | 6 months, 12 months
  DSST (digit symbol substitution test, Wechsler 1981)
Neurocognitive Performance (processing speed 2) | 6 months, 12 months
  TMT-A, -B (Trail-Making-Test, Reitan 1956)
Socialcognitive Performance (affect recognition) | 6 months, 12 months
  PFA (Picture of Facial Affect Test, Ekman & Friesen 1976)
Socialcognitive Performance (theory of mind) | 6 months, 12 months
  MASC (Movie for the Assessment of Social Cognition, Dziobek et al. 2006)
Psychopathology/Symptoms 1 | 6 months, 12 months
  PANSS (Positive and Negative Syndrome Scale, Kay, Fiszbein & Opler 1987)
Psychopathology/Symptoms 2 | 6 months, 12 months
  CDSS (Calgary Depression Rating Scale for Schizophrenia, Addington, Addington & Maticka-Tyndale 1993)
Psychopathology/Symptoms 3 | 6 months, 12 months
  BSI (Brief Symptom Inventory, Derogatis & Melisaratos 1983)
Suicidality | Assessed every 4-6 weeks from date of randomization until 1 year or until discontinuation (whatever came first)
  Incidence of suicide/suicide attempt or severe suicidal crisis (CDSS Item 8 ≥ 2)
Severe symptom worsening | Assessed every 4-6 weeks from date of randomization until 1 year or until discontinuation (whatever came first)
  CGI (Clinical Global Impression Scale Item 2 ≥ 6)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wölwer, Prof. Dr., Principal Investigator — Dept. of Psychiatry and Psychotherapy, University of Düsseldorf
Locations (6):
- Germany (6):
  - Rheinhessen-Fachklinik Alzey, Alzey
  - Vivantes Klinikum Am Urban, Berlin
  - Dept. of Psychiatry and Psychotherapy, University of Bonn, Bonn
  - Dept. of Psychiatry and Psychotherapy, University of Cologne, Cologne
  - Dept. of Psychiatry and Psychotherapy, University of Düsseldorf, Düsseldorf
  - Dept. of Psychiatry and Psychotherapy, University of Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: Yes
Data shall be shared within the German research network ESPRIT (Enhancing Schizophrenia Prevention and Recovery through Innovative Treatments) as well as with other German research networks funded by the BMBF (call "Psychische Erkrankungen").

REFERENCES:
- [Derived] Schuster T, Lowe A, Weide K, Kamp D, Riesbeck M, Bechdolf A, Brockhaus-Dumke A, Hurlemann R, Muthesius A, Klingberg S, Hellmich M, Schmied S, Meyer-Lindenberg A, Wolwer W; ISST study group. Feasibility of six-month outpatient cognitive remediation in schizophrenia: Experience from the randomized controlled integrated social cognition and social skills therapy study. Schizophr Res Cogn. 2023 Apr 27;33:100285. doi: 10.1016/j.scog.2023.100285. eCollection 2023 Sep. PMID 37159610
- [Derived] Wolwer W, Frommann N, Lowe A, Kamp D, Weide K, Bechdolf A, Brockhaus-Dumke A, Hurlemann R, Muthesius A, Klingberg S, Hellmich M, Schmied S, Meyer-Lindenberg A; ISST study group. Efficacy of Integrated Social Cognitive Remediation vs. Neurocognitive Remediation in Improving Functional Outcome in Schizophrenia: Concept and Design of a Multicenter, Single-Blind RCT (The ISST Study). Front Psychiatry. 2022 Jun 21;13:909370. doi: 10.3389/fpsyt.2022.909370. eCollection 2022. PMID 35800017